CLINICAL TRIAL: NCT04104958
Title: Identification of Recent Biomarkers in Polycystic Ovary Syndrome Patients as a Predictors of IVF Outcome
Brief Title: IVF Outcome in Polycystic Ovary Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Engy Mohamed Fikry, Assistant Lecture, Assiut University
Other Study IDs: PCOS IVF
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Enzyme-Linked Immunosorbent Assay; Blotting, Western

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Follicular fluid and granulosa cell collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 (n=50): women (age 20-40year) with PCOS who are diagnosed according to the criteria of the Rotterdam ESHRE/ASRM-sponsored PCOS consensus workshop group (2003), which require two of the following 3 manifestations:
  1. oligo- or anovulation,
  2. clinical and/or biochemical signs of hyperandrogenism (> 2.08 nmol/l),
  3. polycystic ovaries on ultrasound examination (the presence of ≥12 follicles measuring 2-9 mm in diameter and/or ovarian volume > 10 cm)
  Interventions: Genetic: qRTPCR (mRNA level).
- Group 2: Group 2 (n=50): women (age 20-40 year) with male factor infertility.
  Interventions: Genetic: qRTPCR (mRNA level).

INTERVENTIONS:
Genetic: qRTPCR (mRNA level). — RNA extraction and RT-qPCR Protein extraction and western blotting ELISA assay
  Other Names: ELISA; western blot analysis

SUMMARY:
1. To investigate the circulating concentrations of phoenixin and their associations with BMI, the concentrations of sex hormones including (LH), (FSH), (E2), (P4), (TT) and steroid hormones enzyme in PCOS patients.
2. To detect the expression PNX and humanin in women with or without PCOS and to elucidate possible correlations with ovarian reserve and clinical outcomes after IVF-ICSI.
3. To investigate relationship between PNX, humanin expression and PI3K/AKT/mTOR and autophagy pathway as a major signaling mechanism in PCOS for targeting new prognostic and therapeutic markers.
4. The study investigates the correlation between oocyte maturity, fertilization, recent biomarkers and a variety of hormonal parameters in follicular fluid.

DETAILED DESCRIPTION:
* In vitro fertilization (IVF) is an important tool for those couples with difficulty conceiving or maintaining a pregnancy. In the United States, infants conceived with IVF account for approximately 1.6% of live births.
* Polycystic ovary syndrome (PCOS), a highly prevalent gynecological disease, is often characterized by amenorrhea, hirsutism, polycystic ovaries on ultrasound scan, elevated serum luteinizing hormone (LH), low serum follicle-stimulating hormone (FSH), anovulatory infertility, pregnancy and neonatal complications; it is also an important cause of infertility in women of reproductive age because of the associated anovulation. IVF are commonly used for PCOS-associated infertility, there are still some questions regarding the paucity of high quality oocyte, low fertilization, and final pregnancy rate in women with PCOS following IVF.
* Depending on the particular criteria used for diagnosis and the population studied, the prevalence of PCOS has been reported to range from 8% to 13% in women of childbearing age women worldwide.
* Phoenixin was recently discovered using a bioinformatics algorithm which utilized information provided by the Human Genome Project A recently discovered hypothalamic neuropeptide phoenixin is involved in the regulation of the reproductive system, anxiety-related behaviors and pain. Phoenixin acts through its receptor, G protein-coupled receptor 173 (GPR173), to activate the cAMP/PKA pathway leading to the phosphorylation of CREB (pCREB).
* The expression of PNX and GPR173 in HGrC1 by RTPCR and Western blotting. Immunohistochemistry revealed that PNX and GPR173 are present in oocytes, granulosa cells and theca cells at different stages of follicular development in human ovary. GPR173 expression in theca cells increased according to follicle development. Treatment of HGrC1 cells with PNX-14 resulted in a significant upregulation of steroidogenesis enzymes: steroidogenic acute regulatory protein, side-chain cleavage enzyme, aromatase, 3β-HSD, and 17α-OH.These results suggest that PNX expressed in human follicles is possibly involved in folliculogenesis and steroidogenesis.
* In the heart, phoenixin has been shown to decrease myocardial apoptosis by enhancing the expression of the anti-apoptotic factor, Bcl-2 and reducing proapoptotic factors such as Bax, Caspase 3, Cytochrome C and p38 MAPK. Also, these cascades are activated in hearts exposed to PNX during the early reperfusion. Using selective inhibitors of specific targets of cardio protection, such as PI3K and by performing WB analysis of phosphorylated proteins of upstream Akt,, we revealed the involvement of this cascade in PNX-dependent cardio protection. Phoenixin might have induced proliferation in part by reducing apoptosis in GCs via the same mechanism.
* Activation of the phosphatidylinositol 3-kinase (PI3K)/Akt pathway protects against PCOS, which is attributed to prevention of cell apoptosis, facilitation of cell proliferation, induction or prevention of cell autophagy, alleviation of oxidative damage, and adaptation of hypoxia microenvironment.
* PNX may be associated with risk of developing PCOS. They proposed that PNX may provide a connection between multiple pathways contributing to PCOS including androgen action, insulin axis and apoptosis. PNX can serve as a new potential therapeutic target for PCOS patients undergo IVF and improved IVF outcome.
* Humanin is a small neuroprotective peptide identified from cDNA library of AD patient. Since its discovery, humanin has been shown to regulate many biological processes such as apoptosis, cell survival, metabolism, inflammation and oxidative stress. Published evidence suggests that humanin is secreted and expressed in many tissues, including the brain, retinal pigment epithelium, blood vessels, pancreatic beta cell, tumors and testes.
* Published evidence demonstrated the localization and distribution of humanin in human ovarian cells. Strong humanin expression was found in the ovary in multiple types of cells, including granulosa cells, oocytes and stromal cells. Further study revealed that follicular fluid humanin levels were correlated with ovarian reserve markers, and were associated with clinical pregnancy for women undergoing IVF-ICSI.
* Humanin is considered to exert a protective effect against apoptosis and oxidative stress. In preeclampsia, the rate of apoptosis was found to be increased, as a result of the oxidative stress that occurs in placenta.
* It is reported that abnormal insulin signaling is correlated with PCOS (11). IRS-1 is a key factor in insulin signaling pathway which has no kinase activity but its activity is regulated by phosphorylation/dephosphorylation. Serine phosphorylation,of IRS-1 would inhibit IRS-1 activity and block the activation of downstream signaling factors, leading to insulin resistance.
* There were no published data concerning humanin concentrations in pregnancy, especially in PCOS. Our study is the first to provide some expectations for such an association, demonstrating that humanin concentrations are increased in women with PCOS compared to controls.
* Autophagy is a lysosome mediated cellular process to clear misfolded protein, old or damaged organelle in the eukaryotes. Autophagy is an important mechanism to maintain cellular homeostasis and prevent tissue necrosis. Decreased expression of autophagy is associated with poor development of embryo and implantation failure. Moreover, Autophagy is physiologically involved in early normal gestation.
* mTOR is the crosstalk mediator between insulin signaling pathway and autophagy regulation. Insulin sensitivity is positively correlated with autophagy activity in pancreatic β cells, and insulin resistance is a common risk factor for both PCOS and type II diabetes.
* The present study demonstrate that humanin could regulate insulin signaling through IRS-1/mTOR in the hippocampus of APP/SP1 transgenic mice, decrease insulin resistance, improve autophagy in the neuron, decrease Aβ deposition and plaque formation, and improve learning ability and memory. These findings suggest that brain insulin signaling pathway, especially IRS-1/mTOR may be involved in autophagy regulation.
* Humanin treatment could enhance autophagy initiation and autophagy flux and decrease the accumulation of autophagosome to alleviate autophagy malfunction and improved IVF outcome in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* • The diagnosis included donors, male factor infertility and PCOS women.

  * Age ranging from 20 to 40 years

Exclusion Criteria:

* • There were no other etiologies for the PCOS cases, such as congenital adrenal hyperplasia, 21-hydroxylase deficiency, androgen-secreting tumors, Cushing's syndrome, thyroid disease, and hyperprolactinemia.

  * Patients with endometriosis.
  * Patients with history of coronary artery disease, hypertension, liver cirrhosis or hematologic disorders.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: PCOS who are diagnosed according to the criteria of the Rotterdam ESHRE/ASRM-sponsored PCOS consensus workshop group (2003), which require two of the following 3 manifestations:
  1. oligo- or anovulation,
  2. clinical and/or biochemical signs of hyperandrogenism (> 2.08 nmol/l),
  3. polycystic ovaries on ultrasound examination (the presence of ≥12 follicles measuring 2-9 mm in diameter and/or ovarian volume > 10 cm)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Detect difference in expression of phoenixin and humanin in PCOS | Baseline
  Detect difference in expression of phoenixin and humanin markers in follicular fluid and their role in pathogenesis of PCOS.
Assess the link between phoenixin and humanin through the PI3/AKT/mTOR | Baseline
  Assess the link between phoenixin and humanin through the PI3/AKT/mTOR and autophagy signalling pathway that may be considered as a future therapeutic target in PCOS patients to improve IVF outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Mahros Zakhary farag, Professor, Principal Investigator — Faculty of medicin Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao M, Zhou F, Tang L, Zeng Z, Hu S, Wang Y, Ke D, Cheng G, Xia W, Zhang L, Zhu C. Follicular fluid humanin concentration is related to ovarian reserve markers and clinical pregnancy after IVF-ICSI: a pilot study. Reprod Biomed Online. 2019 Jan;38(1):108-117. doi: 10.1016/j.rbmo.2018.11.002. Epub 2018 Nov 23. PMID 30503199
- [Background] Nguyen XP, Nakamura T, Osuka S, Bayasula B, Nakanishi N, Kasahara Y, Muraoka A, Hayashi S, Nagai T, Murase T, Goto M, Iwase A, Kikkawa F. Effect of the neuropeptide phoenixin and its receptor GPR173 during folliculogenesis. Reproduction. 2019 Jul;158(1):25-34. doi: 10.1530/REP-19-0025. PMID 30933929
- [Background] Avagliano L, Terraneo L, Virgili E, Martinelli C, Doi P, Samaja M, Bulfamante GP, Marconi AM. Autophagy in Normal and Abnormal Early Human Pregnancies. Reprod Sci. 2015 Jul;22(7):838-44. doi: 10.1177/1933719114565036. Epub 2014 Dec 28. PMID 25544676
- [Background] Bozdag G, Mumusoglu S, Zengin D, Karabulut E, Yildiz BO. The prevalence and phenotypic features of polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod. 2016 Dec;31(12):2841-2855. doi: 10.1093/humrep/dew218. Epub 2016 Sep 22. PMID 27664216